CLINICAL TRIAL: NCT04885881
Title: The Effectiveness of Ozone (O2-O3) Injections in the Treatment of Myofascial Pain Syndrome: A Prospective Randomized Controlled Study
Brief Title: The Effectiveness of Ozone (O2-O3) Injections in the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Myofascial Pain Syndrome; Myofascial Trigger Point Pain
Keywords: myofascial pain syndrome; trigger point pain; ozone; lidocaine
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone therapy group (Active Comparator): Patients with myofascial pain syndrome receiving ozone injection
  Interventions: Procedure: Ozone therapy
- Lidocaine injection group (Active Comparator): Patients with myofascial pain syndrome receiving lidocaine injection
  Interventions: Procedure: Lidocaine injection group

INTERVENTIONS:
Procedure: Ozone therapy — Patients in the ozone therapy group will be treated with ozone (O2-O3) in a volume of 5 ml and a dose of 10 µg / ml for three consecutive weeks in a weekly session to the most painful trigger point.
  Arms: Ozone therapy group
Procedure: Lidocaine injection group — Patients in the lidocaine injection group will be applied to the most painful trigger point in a volume of 2 ml of 1% lidocaine for three consecutive weeks, once a week.
  Arms: Lidocaine injection group

SUMMARY:
Ozone (O2-O3) has been used as a supportive therapy in various musculoskeletal diseases such as lumbosacral disc herniation, knee osteoarthritis, meniscus injury, shoulder pathologies.The aim of this study is to investigate the effectiveness of ozone (O2-O3) injection applied to the trigger point in the treatment of myofascial pain syndrome.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, controlled trial. Fourty six people who met the inclusion criteria will randomized into two groups of 23 people. The first group will be designated as ozone therapy group and patients in the second group will be designated as the lidocaine injection group. Patients will be evaluated with visuel analog scale (10cm-VAS), Neck Disability Index (NDI), Pain Score (PS) and neck lateral flexion measurement before and after treatment at 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with myofascial pain syndrome according to the criteria defined by Simons et al.
* aged between18-65
* having typical myofascial pain symptoms for at least 3 months

Exclusion Criteria:

* presence of cervical radiculopathy, cervical myelopathy, severe dyscal or bony degeneration
* presence of a history of neck trauma or surgery in the last year
* presence of trigger point injection for myofascial pain syndrome treatment in the last 3 months
* presence of cognitive impairment, malignant hypertension, G6PDH (Glucose 6- Phosphate Dehydrogenase) deficiency, Graves' disease, chronic recurrent pancreatitis attack, severe thrombocytopenia (platelet value <50,000 / microliter), cerebrovascular disease in which bleeding is active
* presence of systemic diseases such as fibromyalgia, inflammatory diseases such as rheumatoid arthritis, polyneuropathy, coagulopathy.
* presence of pregnancy and breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Neck Pain | baseline, change from baseline VAS at 4 and 12 weeks after injection
  Severity of pain was assessed using the standard 10 cm VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | baseline, change from baseline NDI at 4 and 12 after injection
  Neck Disability Index (NDI) is a self-report 10-item questionnaire used to evaluate the effect of neck pain on daily living activities. Each item is scored from 0 to 5. Higher scores of NDI indicate more disability and pain.
Pain Scor (PS) | baseline, change from baseline PS at 4 and 12 weeks after injection
  Pain Scor (PS) measures the severity of pain felt at the trigger point by placing the thumb to the skin covering the muscle containing the trigger point in a perpendicular fashion and exerting pressure until there was whitening of the nail bed.
Range of Motion (ROM) of the neck | baseline, change from baseline ROM at 4 and 12 weeks after injection
  Passive ROM measurements of the neck lateral flexion movements were recorded by a universal goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Korkmaz, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, Department of PMR
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)